CLINICAL TRIAL: NCT02002026
Title: Uterine Artery Ligation to Minimize Blood Loss in Patients With Central Placenta Previa
Brief Title: Uterine Artery Ligation to Decrease Blood Loss With Central Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia Maternity University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Sameer Sanad, Assistant Professor, Minia Maternity University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1150-4666
Record Dates: First submitted 2013-11-18; First posted 2013-12-05 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Placenta Previa Without Hemorrhage
Keywords: placenta previa, uterine artery ligation
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ligation group (Active Comparator): Uterine artery ligation will be done for patients in this group
  Interventions: Procedure: Uterine artery ligation
- Control group (Placebo Comparator): Conventional CS
  Interventions: Procedure: Uterine artery ligation

INTERVENTIONS:
Procedure: Uterine artery ligation — Uterine artery ligation during cesarean section before delivery of the baby

SUMMARY:
This trial will address the effect of uterine artery ligation during Cesarean section in cases with placenta previa to decrease blood loss.

DETAILED DESCRIPTION:
This Study will address the effect of uterine artery ligation prior to fetal delivery during Cesarean section in cases with central placenta previa to guard against postpartum hemorrhage and to minimize blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Placenta previa is diagnosed when the lowest placental edge is located within 5 cm of the internal os at ultrasound
* Symptomatic Placenta previa with at least one episode of bleeding
* Estimated gestational age within 28 to 40 weeks
* Maternal age > 18 years
* Informed consent
* Social affiliation

Exclusion Criteria:

* Premature rupture of membranes
* Severe bleeding.
* Abnormal fetal heart rates.
* Pre-eclampsia, chorioamnionitis, severe chronic renal disease.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in hemoglobin level | hemoglobin level will be done baseline and will be repeated 24 hours after delivery
  Changes in hemoglobin level before and after CS will reflect the amount of blood loss during operation

SECONDARY OUTCOMES:
Degree of uterine contractility. | During CS and within 3 hours after CS

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Sameer, MD, Principal Investigator — Minia Maternity University Hospital
Locations (1):
- Minia Maternity University Hospital, Minya, Minya Governorate, Egypt

REFERENCES:
- [Derived] Sanad AS, Mahran AE, Aboulfotouh ME, Kamel HH, Mohammed HF, Bahaa HA, Elkateeb RR, Abdelazim AG, El-Din MAZ, Shawki HE. The effect of uterine artery ligation in patients with central placenta pevia: a randomized controlled trial. BMC Pregnancy Childbirth. 2018 Aug 29;18(1):351. doi: 10.1186/s12884-018-1989-5. PMID 30157787